CLINICAL TRIAL: NCT07211958
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of Revumenib in Combination With Intensive Chemotherapy in Participants With Newly Diagnosed AML With an NPM1 Mutation
Brief Title: Study of Revumenib in Combination With Intensive Chemotherapy in Newly Diagnosed Acute Myeloid Leukemia (AML) With a NPM1 Mutation
Acronym: REVEAL-ND NPM1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Syndax Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNDX-5613-0710; 2025-522279-27-00 (EU CTIS Number)
Expanded Access: NCT05918913 (No longer available)
Record Dates: First submitted 2025-09-30; First posted 2025-10-08 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Acute Myeloid Leukemias
Keywords: SNDX-5613; Nucleophosmin 1; NPM1; Acute Myeloid Leukemias; AML; Revumenib; Newly diagnosed AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — revumenib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Revumenib + Intensive Chemotherapy (Experimental): Participants will receive revumenib plus an intensive chemotherapy regimen.
  Interventions: Drug: Revumenib; Drug: Intensive Chemotherapy Regimen
- Placebo + Intensive Chemotherapy (Placebo Comparator): Participants will receive placebo plus an intensive chemotherapy regimen.
  Interventions: Drug: Placebo; Drug: Intensive Chemotherapy Regimen

INTERVENTIONS:
Drug: Revumenib — Participants will receive revumenib orally.
  Other Names: SNDX-5613
  Arms: Revumenib + Intensive Chemotherapy
Drug: Placebo — Participants will receive placebo (non-active agent) orally.
  Arms: Placebo + Intensive Chemotherapy
Drug: Intensive Chemotherapy Regimen — Participants will receive an intensive chemotherapy regimen of cytarabine and daunorubicin by intravenous (IV) infusion.

SUMMARY:
The purpose of this study is to assess if adding revumenib to standard chemotherapy improves outcomes in participants with AML with certain genetic mutations compared to chemotherapy alone. The study will also assess the safety of adding revumenib to chemotherapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants must have newly diagnosed and previously untreated AML and be candidates for intensive chemotherapy.
* Presence of an NPM1 mutation.
* Eastern Cooperative Oncology Group performance status ≤2 (≤1 if >65 years old); Karnofsky or Lansky ≥40.
* Have a life expectancy of ≥3 months as judged by the Investigator.
* Negative serum pregnancy test.
* Adequate liver, kidney, and cardiac function.

Key Exclusion Criteria:

* Diagnosis of active acute promyelocytic leukemia.
* Active central nervous system disease.
* Fridericia's corrected QT interval (QTcF) >450 milliseconds at screening, diagnosis or suspicion of Long QT syndrome or family history of Long QT syndrome.
* Any gastrointestinal (GI) issue of the upper GI tract likely to affect oral drug absorption or ingestion.
* Any concurrent malignancy requiring active therapy (except breast or prostate cancer stable on or responding to endocrine therapy).
* Inability to swallow oral medication.
* Pregnant or nursing females.
* Participant has known active or chronic hepatitis B or active hepatitis C (HCV) infection or human immunodeficiency virus (HIV)-positive with detectable viral load.

Note: Additional inclusion/exclusion criteria may apply, per protocol.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 468 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Event Free Survival | Up to 2 years
Measurable Residual Disease Complete Remission Rate | Up to 2 years

SECONDARY OUTCOMES:
Overall Survival | Up to 5 years
Rate of Complete Remission | Up to 2 years
Overall Response Rate | Up to 2 years
Duration of Complete Remission | Up to 2 years
Duration of Composite Complete Remission | Up to 2 years
Duration of Response | Up to 2 years
Number of Participants with a Treatment-emergent Adverse Event | Up to 2 years
Change from Baseline in Patient-reported Fatigue Questionnaire Scores | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (3):
- Georgia (2):
  - Clinical Trial Site, Batumi, Adjara
  - Clinical Trial Site, Tbilisi
- Clinical Trial Site, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No